CLINICAL TRIAL: NCT05045183
Title: A 16-Day, Single-Center, Randomized, Comparator-Controlled Study to Assess Wound Healing Efficacies of Different Clean, Treat, and Protect Wound Care Regimens Compared to Standard of Care and Untreated
Brief Title: A Study to Assess Wound Healing Efficacies of Different Clean, Treat, and Protect Wound Care Regimens Compared to Standard of Care and Untreated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCSTOH003808; CCSTOH003808 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2022-10

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment A: Uncovered Wound (Negative Control) (No Intervention): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, no treatment will be applied as the wound will be kept uncovered as a negative control.
- Treatment B: Standard of Care (SoC) Adhesive Bandage (Active Comparator): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, SoC adhesive bandage will be applied. This treatment will be changed daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Device: SoC Adhesive Bandage
- Treatment C: Antibiotic Ointment (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, antibiotic ointment will be applied. This treatment will be applied daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Drug: Antibiotic Ointment
- Treatment D: Antibiotic Ointment Plus SoC Adhesive Bandage (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, antibiotic ointment plus SoC adhesive bandage will be applied. This treatment will be applied and changed daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Device: SoC Adhesive Bandage; Drug: Antibiotic Ointment
- Treatment E: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, antiseptic wash plus antibiotic ointment plus SoC adhesive bandage will be applied. This treatment will be applied and changed daily from Day 0 through Day 2 and all wound sites will be uncovered after Day 3 to Day 16 for assessments.
  Interventions: Device: SoC Adhesive Bandage; Drug: Antibiotic Ointment; Drug: Antiseptic Wash
- Treatment F: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, antiseptic wash plus antibiotic ointment plus SoC adhesive bandage will be applied. This treatment will be applied and changed daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Device: SoC Adhesive Bandage; Drug: Antibiotic Ointment; Drug: Antiseptic Wash
- Treatment G: Hydrocolloid Pad (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, hydrocolloid pad will be applied. This treatment will be changed daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Device: Hydrocolloid Pad
- Treatment H: Hydrocolloid Pad (Experimental): Minor wounds will be created on participant's forearms (four per arm) by a certified laser specialist. On the randomized wound site, hydrocolloid pad will be applied. This treatment will be changed daily from Day 1 through Day 6 and all wound sites will be uncovered from Day 7 to Day 16 for assessments.
  Interventions: Device: Hydrocolloid Pad

INTERVENTIONS:
Device: SoC Adhesive Bandage — On the randomized wound site, a SoC adhesive bandage will be applied.
  Arms: Treatment B: Standard of Care (SoC) Adhesive Bandage; Treatment D: Antibiotic Ointment Plus SoC Adhesive Bandage; Treatment E: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage; Treatment F: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage
Drug: Antibiotic Ointment — On the randomized wound site, a antibiotic ointment will be applied.
  Arms: Treatment C: Antibiotic Ointment; Treatment D: Antibiotic Ointment Plus SoC Adhesive Bandage; Treatment E: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage; Treatment F: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage
Drug: Antiseptic Wash — On the randomized wound site, a antiseptic wash will be applied.
  Arms: Treatment E: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage; Treatment F: Antiseptic Wash Plus Antibiotic Ointment Plus SoC Adhesive Bandage
Device: Hydrocolloid Pad — On the randomized wound site, hydrocolloid pad will be applied.
  Arms: Treatment G: Hydrocolloid Pad; Treatment H: Hydrocolloid Pad

SUMMARY:
The purpose of this study is to evaluate the healing rates of wounds treated with various wound care regimens including antiseptic wound wash, topical antibiotic treatment, adhesive bandages, and/or hydrocolloid bandages.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I to III
* Uniform skin color on both volar forearms
* Generally in good health based on medical history reported by the participant, and as verified by the Principal Investigator (PI) assessment and brief interview of medical history
* Able to read, write, speak, and understand English
* Individual must be able to understand the nature, risk, and relevance of the study
* Individual has signed the Consent for Photograph Release and informed consent document (ICD) including Health Insurance Portability and Accountability Act (HIPAA) disclosure after the nature of the study has been fully explained
* Willing to undergo topical anesthetic and laser wound treatment on the volar forearms
* Individual must agree to attend all required study visits, cooperate/follow all study instructions, and participate with all the procedures for the duration of the study and return to the clinical site for all scheduled visits as required by the investigator
* Willing to wear long sleeves when going outdoors during the study to protect the test areas from exposure to sunlight. Individuals must agree to avoid exposing their forearms to sunlight (including tanning booths) throughout the entire study period
* Individual must agree not to immerse their bandages in water for the duration of the study. Participants will only be allowed to shower during the course of the study (no swimming, baths, hot tubs, Et cetera [etc.]) Individuals must agree not to shower within 2 hours prior to each scheduled visit
* Individuals must agree not to use lotions, creams, moisturizers, cosmetics, or sunscreens on their forearms (sites of wounds) for the entire duration of the study
* Individuals must agree to refrain from the use of any daily cleanser or washoff products other than the auxiliary cleanser that will be provided at screening (that is, [Day -7 to Day -3]), for use on forearms throughout the study

Exclusion Criteria:

* Has known allergies, hypersensitivity, or adverse reactions to anesthetics, adhesive bandages, latex, wound treatment products, or any component/ingredient present in the investigational products (IPs)/auxiliary/ancillary products
* Has a known history of a blood-clotting disorder, cardiovascular, hepatic, or kidney disease
* Presents with a known history of keloid or hypertrophic scar formation, cracked or excoriated skin, clinical infected skin lesions, or other skin problems that would in the opinion of the PI or Study Physician, confound the study results, increase risk to the participant, or interfere with study evaluations (example, active psoriasis anywhere on the body, seborrheic dermatitis, atopic dermatitis, other skin dermatoses, etc.)
* Has excessive hair, acne, scars, pigmentation, tattoos, or friable skin on either volar forearm that could interfere with evaluations or study procedures (at the discretion of the PI)
* Has a known history of severe systemic immune system disorders such as Systemic Lupus Erythematosus (SLE), Rheumatoid Arthritis (RA), Scleroderma, chronic connective tissue disorders, Poly Arteritis Nodosa, or immunodeficiency, including human immunodeficiency viruses (HIV) infection
* Has a history of a confirmed Coronavirus Disease 2019 (COVID-19) infection within 30 days prior to Visit 1
* Has had contact with a COVID-19 infected person within 14 days prior to Visit 1
* Individual or a member of the individual's household who has traveled internationally within 14 days prior to Visit 1
* Has experienced any of the following self-reported symptoms of COVID-19 within 2 weeks prior to the study visit: a) Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches) conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness; b) Temperature greater than or equal to (>=) 37.2 degree Celsius (°C)/99.5 degree Fahrenheit (°F), measured; c) Use of fever reducers within 2 days prior to each on-site study visit
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Has self-reported uncontrolled chronic diseases such as hypertension, hyperthyroidism, hypothyroidism, or active or recently treated (within 1 year) skin cancer, or those in known poor nutritional status
* Is taking a medication that would mask an Adverse Event (AE), confound the study results, or alter or compromise the bleeding/healing process including: a) Antibiotics, oral corticosteroids, immunosuppressive agents, anti-coagulants, antiplatelet drugs, cytotoxic agents, continuous aspirin therapy, chemotherapy, or daily medications for chronic asthma, within 1 month before Visit 1; b) Non-steroidal anti-inflammatory drugs or steroidal drugs within 5 days before Visit 1. Low dose aspirin (81 milligrams [mg] per day) is allowed; c) Antihistamines within 2 weeks before Visit 1
* Is self-reported to be pregnant, lactating or planning to become pregnant during the study
* Has taken/used (oral or topical) vitamin A derivatives such as Accutane, isotretinoin, or retinoic acid within the past 1 year, or using topical Vitamin A derivatives on the forearms in the 3 weeks prior to Visit 1.
* Has used topical leave-on products on the volar forearms within 1 week prior to Visit 1
* Is participating or has participated in 1) any clinical trial involving a topical or systemic investigational drug within 30 days prior to Visit 1 or 2) any other clinical study within 10 days prior to Visit 1
* Has a body mass index (BMI) above 35 on the BMI scale. BMI will be calculated using height and weight measurements obtained by trained study personnel
* Is self-reported to be an alcohol or drug abuser, or with any other known severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the PI, would make the participant inappropriate for entry into this study
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor
* Has a relative, partner, or staff of any clinical research site personnel, or either is or lives with someone who is a current employee of any company that makes or markets adhesive bandages or first aid products
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study or viewed by the PI as not being able to complete the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Composite Healing Score | Day 0 through Day 7
  Composite healing score will be calculated from clinical grading of wound healing parameters as (general wound appearance score plus [+] smoothness score + epithelial confluence score) minus [-] (erythema score + edema score + crusting/scabbing score). Composite healing score on a 25-point scale (-12 [no healing] to +12 [towards healing]) is indicative of extent of wound healing and will be calculated for each wound site at each evaluation day.
Composite Healing Score | Day 16
  Composite healing score will be calculated from clinical grading of wound healing parameters as (general wound appearance score + smoothness score + epithelial confluence score) - (erythema score + edema score + crusting/scabbing score). Composite healing score on a 25-point scale (-12 [no healing] to +12 [towards healing]) is indicative of extent of wound healing and will be calculated for each wound site at each evaluation day.

SECONDARY OUTCOMES:
Clinical Grading of Wound Healing of Erythema | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of erythema will be reported. It will be evaluated on a scale of 0 to 4 with 0=none/absent, 1=mild, 2=moderate, 3=marked, and 4=severe, with higher scores indicating a worse outcome.
Clinical Grading of Wound Healing of Edema | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of edema will be reported. It will be evaluated on a scale of 0 to 4 with 0=none/absent, 1=mild, 2=moderate, 3=marked, and 4=severe, with higher scores indicating a worse outcome.
Clinical Grading of Wound Healing of General Wound Appearance | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of general wound appearance will be reported. It is evaluated on a scale from 0 to 4 with 0=poor, 1=fair, 2=good, 3=very good, 4=excellent with higher scores indicating a better outcome.
Clinical Grading of Wound Healing of Smoothness | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of smoothness of popped pimple as assessed by trained grader will be reported. It will be evaluated on a scale of 0 to 4 with 0=rough, uneven wound, 1=mild smoothness, 2=moderate smoothness, 3=extensive smoothness, and 4=complete smooth, even wound, with higher scores indicating a better outcome.
Clinical Grading of Wound Healing of Epithelial Confluence | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of epithelial confluence will be reported. It will be evaluated on a scale from 0 to 4 with 0=none (no epithelial coverage), 1=slight (up to 30 percent [%]), 2=moderate (31% to 60%), 3=extensive (61% to 90%), and 4=almost complete or complete (91% to 100%, covered with a full layer of new epithelial growth), with higher scores indicating a better outcome.
Clinical Grading of Wound Healing of Crusting/Scabbing | Day 0 through Day 7, Day 16
  Clinical grading of wound healing of crusting/scabbing will be reported. It will be evaluated on a scale of 0 to 4 with 0=none, 1=slight (up to 30%), 2=moderate (31% to 60%), 3=extensive (61% to 90%), and 4=almost complete or complete (91% to 100%), with higher scores indicating a worse outcome.
Wound Healing Process Assessment Score | Day 16
  Wound healing process assessment of each test site will be performed and a score of "0" or "1" will be assigned where 0=primary healing (the wound heals by primary epithelial tissue), and 1=secondary healing (the wound heals through the stage of formation of connective tissue).
Painful Score with Arm Resting by Side (Participant's Self-assessment Questionnaire) | Day 0 through Day 7, Day 16
  Painful score with arm resting by side based on participants self-assessment questionnaire score (question 1) will be reported. Participants will be asked to rate each wound for pain/soreness in resting position as score from 0 (no pain) to 10 (severe pain).
Pain Duration with Arm Resting by Side (Participant's Self-assessment Questionnaire) | Day 0 through Day 7, Day 16
  Participants will be asked to rate the pain as either brief, periodic, or constant in arm resting position with the Self-assessment questionnaire (question 2).
Painful Score with Arm in Normal Motion (Participant's Self-assessment Questionnaire) | Day 0 through Day 7, Day 16
  Painful Score based on participants self-assessment questionnaire score (question 3) will be reported. Participants will be asked to rate each wound for pain/soreness in normal position as score from 0 (no pain) to 10 (severe pain).
Pain Duration with Arm in Normal Motion (Participant's Self-assessment Questionnaire) | Day 0 through Day 7, Day 16
  Participants will be asked to rate the pain as either brief, periodic, or constant in arm normal motion with the Self-Assessment Questionnaire (question 4).
Itchy Score of Wound Site (Participant's Self-assessment Questionnaire) | Day 0 through Day 7, Day 16
  Itchy score based on participants self-assessment questionnaire score (question 5) will be reported. Participants will be asked to rate each wound for itchiness as score from 0 (no itch) to 10 (severe itch).

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Emmerich, Ph.D., Principal Investigator — SGS Stephens, Inc. Dallas Research Center
Locations (1):
- SGS Stephens, Inc. Dallas Research Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Mancini AJ, Sookdeo-Drost S, Madison KC, Smoller BR, Lane AT. Semipermeable dressings improve epidermal barrier function in premature infants. Pediatr Res. 1994 Sep;36(3):306-14. doi: 10.1203/00006450-199409000-00007. PMID 7808826
- [Background] WINTER GD. Formation of the scab and the rate of epithelization of superficial wounds in the skin of the young domestic pig. Nature. 1962 Jan 20;193:293-4. doi: 10.1038/193293a0. No abstract available. PMID 14007593
- [Background] Winter GD. Some factors affecting skin and wound healing. J Tissue Viability. 2006 May;16(2):20-3. doi: 10.1016/s0965-206x(06)62006-8. PMID 16752710
- [Background] Bernard DB. Chapter 41: Minor Burns, Sunburns, and Wounds. In Krinsky DL, Ferreri SP, and Hemstreet B., et al., Handbook of nonprescription drugs: An interactive approach to self-care (19th ed.) Washington, DC: American Pharmacists Association. doi:https://doi-org.jerome.stjohns.edu/10.21019/9781582122656.ch41
- [Background] Cuts and scrapes: First aid. (2019, October 29). Retrieved January 22, 2021, from https://www.mayoclinic.org/first-aid/first-aid-cuts/basics/art-20056711
- [Background] Trookman NS, Rizer RL, Weber T. Treatment of minor wounds from dermatologic procedures: a comparison of three topical wound care ointments using a laser wound model. J Am Acad Dermatol. 2011 Mar;64(3 Suppl):S8-15. doi: 10.1016/j.jaad.2010.11.011. Epub 2011 Jan 17. PMID 21247665
- [Background] NIH Publication No. 98-4083 (1998, September). Adapted from Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults: The Evidence Report. Retrieved from URL. https://www.nhlbi.nih.gov/health/educational/lose_wt/BMI/bmi_tbl.htm. 22 May 2019.
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSTOH003808&attachmentIdentifier=2a69ca5a-f229-44da-8dc3-2fb7a414144e&fileName=CCSTOH003808_Summary_CSR_Final_Version_1.0__13_Oct_2002__Redacted.pdf&versionIdentifier=